CLINICAL TRIAL: NCT00214448
Title: Reproducibility of the GeneTrait™ CGH Microarray System DX Using Whole Blood Samples
Brief Title: Reproducibility of the Array-Based Comparative Genomic Hybridization (aCGH) System Using Whole Blood Samples
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Abbott Molecular (Industry)
Other Study IDs: 05-801
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2005-09

CONDITIONS: Genetic Disorders
Keywords: Multiple genetic conditions will be studied
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The objective of this study is to validate the performance characteristics of the GeneTrait CGH Microarray System DX. Reproducibility among sites, lots, and operators will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to donate at least 10 mL of whole blood
* Must be able to provide consent, or parental consent and patient assent (if applicable)
* Must be currently followed as a patient of a genetic clinic or counselor at one of the recruiting sites
* Must have at least one chromosomal change that is detectable by the GeneTrait CGH Microarray System DX as determined by karyotype and/or fluorescence in situ hybridization (FISH) analysis (within any of the 73 critical regions)

Exclusion Criteria:

* Unable to donate at least 10 mL of whole blood
* Unable to provide consent, or parental consent and patient assent (if applicable)
* Not currently followed as a patient of a genetic clinic or counselor at one of the recruiting sites
* Does not have at least one chromosomal change that is detectable by the GeneTrait CGH Microarray System DX as determined by karyotype and/or FISH analysis (within any of the 73 critical regions)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4